CLINICAL TRIAL: NCT05075187
Title: Epidemiological Study in FRONtoTemporal Dementia
Acronym: EFRONT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: EFRONT 05-2021
Record Dates: First submitted 2021-09-30; First posted 2021-10-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed with Frontotemporal Dementia: Participants diagnosed with Frontotemporal Dementia
  Interventions: Diagnostic Test: Genetic Screening

INTERVENTIONS:
Diagnostic Test: Genetic Screening — Blood samples will be collected from clinically diagnosed or suspected FTD patients and will be analysed for a broad range of pathogenic variants in genes associated with FTD.

SUMMARY:
An international, multicenter, epidemiological observational study aims to investigate the prevalence of genetic etiologies in patients diagnosed with FTD or clinically suspected for FTD.

DETAILED DESCRIPTION:
Frontotemporal dementia (FTD) is a genetically and pathologically heterogeneous neurodegenerative disease caused by the loss or damage of nerve cells in the brain's frontal and temporal lobes. This leads to abnormalities in behaviour, personality, and language comprehension problems. Also, people with FTD show movement disorders like tremor, rigidity, difficulty in coordination, muscle spasms and weakness. FTD's etiology is sporadic or heritable. Sixty to 70% of FTD cases are sporadic, while 30 to 40% are inherited (familial aggregation). For this study, blood samples were collected from clinically diagnosed or suspected FTD patients and were analysed for a broad range of pathogenic variants in genes associated with FTD. The scientific insights acquired from this study will help identify novel therapeutic targets and develop/ investigate potential disease-modifying drugs.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, which includes reference to the genetic testing, is obtained from the participant/legal guardian
* The participant is aged between 25 to 85 years
* The participant is diagnosed with Frontotemporal dementia (FTD) or has signs or symptoms of FTD

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with Frontotemporal Dementia (FTD) and participants clinically suspected for FTD
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the prevalence of genetic etiologies in FTD by genotyping FTD participants/ FTD suspected participants | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Ph.D, Principal Investigator — Centogene GmbH
Locations (37):
- Belgium (2):
  - AZ Damiaan, Ostend, West Flanders
  - CHU de Liege, Liège
- Germany (11):
  - Hanau Hospital, Hanau, Hesse
  - Gertrudis Klinik, Leun, Hesse
  - University Hospital Dresden, Dresden, Saxony
  - University Medical Center Hamburg Eppendorf, Hamburg, Schleswig-Holstein
  - University of Lübeck, Lübeck, Schleswig-Holstein
  - RWTH Aachen University, Aachen
  - Hochtaunus-Kliniken gGmbH, Bad Homburg
  - AGZ of Charite Universitätsmedizin Berlin, Berlin
  - University Hospital Cologne, Cologne
  - Asklepios Klinik Nord - Ochsenzoll, Hamburg
  - University Hospital Rostock, Rostock
- Greece (2):
  - Mediterraneo Hospital, Athens
  - University of Ioannina, Ioannina
- Italy (4):
  - Università degli studi Gabriele D'Annunzio Chieti-Pescara, Chieti
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda USL-IRCCS of Reggio Emilia, Reggio Emilia
- Portugal (6):
  - Hospital Garcia de Orta, Almada
  - Unidade Psiquiatrica Privada de Coimbra, Coimbra
  - Hospital da Senhora da Oliveira Guimaraes, Guimarães
  - Hospital Beatriz Ângelo, Loures
  - Hospital Pedro Hispano, Matosinhos Municipality
  - CNS - campus neurológico Torres Vedras, Torres Vedras
- Spain (6):
  - Hospital Universitari vall D´hebron, Barcelona
  - Universitary Hospital La Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Marqués de Valdecilla University Hospital, Santander
- Turkey (Türkiye) (6):
  - Baskent University, Ankara
  - Hacettepe University, Ankara
  - Koç University Hospital, Istanbul
  - Istanbul University, Istanbul
  - Bezmialem Vakif University, Istanbul
  - Izmir Economy University Medikalpark Hospital, Izmir